CLINICAL TRIAL: NCT04109144
Title: Fresh Frozen Plasma as a Substitute for Albumin in Patients Receiving a Large Volume Paracentesis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI confirmed that while coordination and planning was conducted upon IRB approval, no participants were enrolled into the study
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-10354
Record Dates: First submitted 2019-09-25; First posted 2019-09-30 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Liver Cirrhosis; Ascites Hepatic
Keywords: Paracentesis; Albumin; Plasma
MeSH Terms: conditions — Liver Cirrhosis | interventions — Albumins

STUDY DESIGN:
Intervention Model Description: single arm, single center, investigator initiated, prospective pilot clinical trial study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Large Volume Paracentesis (LVP) with Fresh Frozen Plasma (FFP) (Experimental): All participants who are scheduled for a LVP and meet the eligibility criteria will be monitored for 3 consecutive periods. At the second drainage participants will receive 2 units, or about 500 ccs, of fresh frozen plasma intravenously, plus 1 bottle, or 50 ccs, of 25% albumin if more than 4 liters of fluid are removed
  Interventions: Biological: Fresh Frozen Plasma (FFP); Procedure: Large Volume Paracentesis (LVP)
- Large Volume Paracentesis (LVP) with Albumin (Active Comparator): All participants who are scheduled for a LVP and meet the eligibility criteria will be monitored for 3 consecutive periods. At the first and third drainage participants will receive 1 bottle, or 50 ccs, of 25% albumin intravenously for every two liters of fluid removed
  Interventions: Biological: Albumin; Procedure: Large Volume Paracentesis (LVP)

INTERVENTIONS:
Biological: Fresh Frozen Plasma (FFP) — FFP will be used as a substitute for albumin during the 2nd of 3 total paracentesis being monitored
  Arms: Large Volume Paracentesis (LVP) with Fresh Frozen Plasma (FFP)
Biological: Albumin — Albumin will be used during the 1st and 3rd paracentesis
  Arms: Large Volume Paracentesis (LVP) with Albumin
Procedure: Large Volume Paracentesis (LVP) — All participants who have this procedure, meet eligibility criteria and who consent

SUMMARY:
Large volume paracentesis (LVP) with albumin administration is the standard of care for patients with refractory ascites complicating end-stage liver disease. However, the use of albumin is frequently limited due to expense and occasional short supply. The goal of this study is to determine if the administration of Fresh Frozen Plasma (FFP) during large volume paracentesis is effective in lowering plasma renin activity by 25% compared to baseline.

DETAILED DESCRIPTION:
There will be three periods of this study, one for each of three consecutive routine large volume paracenteses. The length of the study will be 6 days post paracentesis for each period, for a total of 3 periods. The interval between successive LVP's will be determined by patients' need. In order to ensure follow up on Day 6, Day 1 will be restricted to a Tuesday, Wednesday, Thursday, or Friday.

All participants will be monitored for 3 consecutive routine large volume paracenteses. The 3 periods (LVP's) of this study will differ in administration of volume replacement solution. First LVP will be with intravenous albumin (12.5gm 25% Human Albumin for every 2 liters removed), 2nd LVP with administration 1 unit of FFP for every 2 liters removed for the first 4 liters followed by 12.5gm 25% albumin for every subsequent 2 liters removed, and 3rd LVP again with administration of intravenous albumin. The first LVP serves as the study entry time period and also as a control period for the same patient. The second LVP is to test the new intervention with FFP. The third LVP is included so that we can monitor the patient's status.

Albumin or FFP administration:

Albumin administration:

50ml of 25% albumin for every 2L removed

FFP administration:

2 units of FFP for the first 4L removed followed by 50ml of 25% albumin for every additional 2L removed FFP will be supplied by the Blood Bank and albumin from the pharmacy at Montefiore Medical Center.

Details for each study period:

1. st Period: Day 1: Enrollment, baseline pre-LVP laboratory testing and measurements, and large volume paracentesis with administration of albumin Day 6: Laboratory testing and measurements
2. nd Period: Day 1: pre-LVP baseline labs and measurements, LVP with FFP administration Day 6: Laboratory testing and measurements
3. rd Period: Day 1: pre-LVP baseline labs and measurements, LVP with albumin administration Day 6: Laboratory testing and measurements

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Cirrhosis of the liver based on biopsy or clinical and radiographic criteria
3. Ability to provide informed consent (Grade 0 to 1 HE)
4. Grade 3 ascites or refractory ascites
5. Ascites requiring frequent large volume paracentesis of at least 5 liters at least once a month
6. No diuretic use
7. INR > 1.7, <2.5

Exclusion Criteria:

1. Inability to obtain informed consent
2. Age less than 18
3. Hepatic Encephalopathy Grade > 1 as defined by the presence of an impaired mental status or the presence of asterixis
4. Septic shock
5. Active infection
6. Respiratory failure
7. Heart failure with reduced ejection fraction of ≤ 50%
8. Moderate or severe pulmonary hypertension
9. History of stroke
10. Unstable coronary artery disease
11. Chronic kidney disease (GFR <60)
12. GI bleed within 2 weeks
13. Any licorice within 2 weeks of starting the study
14. Any Beta Blocker use within the last 2 weeks
15. Any diuretic use within 2 weeks
16. Absence of paracentesis within 2 weeks
17. Absence of volume expanders within 2 weeks
18. INR > 1.7
19. Pregnancy - pregnancy test will be administered for all female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in plasma renin activity (PRA) post paracentesis | 6 Days
  Efficacy of LVP with FFP will be measured as the change of plasma renin activity (PRA) from Day 1 to Day 6 during the 2nd LVP with FFP. We hypothesize that FFP will reduce the PRA by 25% from Day 1 to Day 6.

SECONDARY OUTCOMES:
Occurrence of post-paracentesis circulatory dysfunction (PPCD) | 6 days
  We hypothesize that the PPCD incidence will reduce in the 2nd LVP with FFP in comparison to the 1st LVP with albumin.
Safety: Adverse Events (AE) | 6 days
  We hypothesize that the overall adverse events (including PPCD incidence) will be reduced in the 2nd LVP with FFP in comparison to the 1st LVP with albumin. AE's will be summarized by presenting the number and percentages of patients having any AE.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Sigal, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No
Data collected during the study will only be shared with researchers that have been IRB approved as key-personnel on the study protocol.